CLINICAL TRIAL: NCT00596453
Title: Impact of Antibiotic Treatment on PSA Variability
Brief Title: Impact of Antibiotic Treatment on Prostate-Specific Antigen (PSA) Variability
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit enough patients
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: NA_00010549
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-11

CONDITIONS: Prostate Infections
Keywords: Prostate Specific Antigen (PSA); Elevated Prostate Specific Antigen (PSA)
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Ciprofloxacin hydrochloride (Experimental)
  Interventions: Drug: Ciprofloxacin hydrochloride

INTERVENTIONS:
Drug: Ciprofloxacin hydrochloride — 250 mg Ciprofloxacin hydrochloride twice a day for 14 days
  Arms: Ciprofloxacin hydrochloride
Drug: Placebo — Placebo twice a day for 14 days
  Arms: Placebo

SUMMARY:
Ciprofloxacin hydrochloride has been approved by the Food and Drug Administration (FDA) for the treatment of mild to moderate infections, including prostate infections. It has been suggested that antibiotic treatment influences PSA levels due to the fact that an increase in PSA levels may be caused by inflammation or swelling of the prostate. Antibiotics are used to treat such inflammatory conditions. However, it has not been proven that antibiotics can be used to lower PSA. This research is being done to see if treatment with the antibiotic Ciprofloxacin hydrochloride affects the Prostate-Specific Antigen (PSA) blood test. This study may also help doctors in deciding which patients need a prostate biopsy.

DETAILED DESCRIPTION:
This study is directed towards men who have been referred to the Urology clinic at the Johns Hopkins Outpatient Center in Baltimore, MD. If a patient fits the eligibility criteria and signs a consent form, the patient will have his blood drawn for the first PSA measurement. The patient must return to the Johns Hopkins Outpatient Center one week later for a second PSA measurement. The patient will be randomized to receive treatment with placebo or Ciprofloxacin hydrochloride for 14 days. The patient must return to the Johns Hopkins Outpatient Center at the end of the treatment cycle for the third PSA measurement. The patient will return one week later for his biopsy and fourth PSA measurement.

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient of Johns Hopkins Urology Outpatient Clinic
* Must have an elevated PSA (> 2.5 ng/mL) and be selected on the basis of a serum PSA evaluation for Transrectal Ultrasound (TRUS)/biopsy
* Must be able to understand and willing to adhere to the study protocol
* Must be willing to take the antibiotic or placebo for two weeks prior to the biopsy and agree to have the biopsy regardless of the change in PSA

Exclusion Criteria:

* Abnormal digital rectal examination
* Anyone currently being treated or who have been treated for any prostatic diseases (prostatitis, prostate Benign Prostatic Hyperplasia (BPH) surgery, prostate cancer) or urinary tract infection in the past
* Anyone taking medications that are likely to alter serum PSA concentration (specifically, androgen steroid hormones, antiandrogens, finasteride, Leutinizing Hormone Releasing Hormone (LHRH) analogues)
* Anyone unwilling to sign the informed consent or who are unlikely to adhere to the study protocol
* Anyone with a known allergy to fluoroquinolone antibiotics
* Anyone on blood thinning medication (Coumadin)
* Anyone taking Tizanidine
* Anyone with a history of seizures or cerebral arteriosclerosis
* Anyone who has taken an antibiotic medication within the past two weeks

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Misop Han, M.D., M.S., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital Outpatient Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants were enrolled but were removed prior to arm/group assignment. One participant was not eligible for the study and the other two participants changed their minds about being part of the research study.
Period: Overall Study
Arm/Group | Placebo | Ciprofloxacin Hydrochloride
Started | 13 | 15
Completed | 12 | 12
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ciprofloxacin Hydrochloride | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 3 | 7 | 10
Age, Continuous [Mean (Full Range); unit: years] | 58.46 [44 to 72] | 62.73 [47 to 71] | 60.75 [44 to 72]
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 15 | 28
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: PSA Levels (Change in PSA Levels With and Without Antibiotics Therapy)
Description: We took 4 Prostate Specific Antigen (PSA, ng/mL) measurements per participant. The first PSA test was performed at enrollment. The second PSA test was performed 7 days (+/-3 days) later. Then the participants took the Placebo or Cipro for 14 days. The participants returned for their 3rd PSA test upon completion of the Placebo or Cipro. The final PSA test was performed 7 days (+/-3 days) after the 3rd test.
  We planned to compare the differences between the first two PSA tests and the last two PSA tests in the Placebo vs Cipro groups.
Time Frame: 1 month post enrollment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Ciprofloxacin Hydrochloride
Number analyzed (Participants) | 13 | 15
ng/mL | 1.23 (0.6) | 0.52 (0.59)

ADVERSE EVENTS:
Arm/Group | Placebo | Ciprofloxacin Hydrochloride
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 1/13 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Ciprofloxacin Hydrochloride (N=15)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes